CLINICAL TRIAL: NCT02590224
Title: Ferrous Bis-glycinate Versus Ferrous Glycine Sulfate for the Treatment of Iron Deficiency Anemia During Pregnancy
Brief Title: The Effect of Iron Deficiency Anemia During Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDA
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferroglycine sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferrous bis-glycinate group (Active Comparator): The patients will receive oral ferrous bis-glycinate fully reacted amino acid 27 mg tablets (Pharaferro 27 tablets) once daily for eight consecutive weeks.
  Interventions: Drug: Ferrous bis-glycinate
- Ferrous glycine sulphate group (Active Comparator): The patients will receive 567.6 mg of ferrous glycine sulphate capsules (Ferrosanol duodenale capsules, Schwarz) once daily for eight consecutive weeks.
  Interventions: Drug: Ferrous glycine sulphate

INTERVENTIONS:
Drug: Ferrous bis-glycinate
  Arms: Ferrous bis-glycinate group
Drug: Ferrous glycine sulphate
  Arms: Ferrous glycine sulphate group

SUMMARY:
Iron deficiency anemia during pregnancy is a significant worldwide health problem, affecting 22% of pregnant women in industrialized countries and 52% in non-industrialized countries. Iron deficiency anemia during pregnancy is associated with increased maternal as well as fetal morbidity, including prematurity, low birth-weight and perinatal and infant loss. Therefore, routine iron supplementation during the second half of pregnancy has been recommended once daily. Others, however, support a selective iron supplementation only for women with iron deficiency anemia, in order to avoid the increased risk of haemoconcentration associated with routine iron supplementation. Unfortunately, compliance to either iron-supplementation programs, especially among pregnant women, is poor, due in part to the side effects associated with these preparations.

Currently, there are many iron preparations available containing different types of iron salts, including ferrous sulfate, ferrous fumarate, ferrous ascorbate but common adverse drug reactions found with these preparations are mainly gastrointestinal intolerance like nausea, vomiting, constipation, diarrhea, abdominal pain, while ferrous bis-glycinate (fully reacted chelated amino acid form of iron) rarely make complication.

Product resulting from the reaction of a metal ion from a soluble salt with amino acids to form coordinate covalent bonds, the resulting molecule is called as chelate and chemical bonding process is called chelation. Ferrous bis-glycinate is highly stable and totally nutritionally functional chelate it is an amino acid fully reacted chelate which is formed by the binding of two molecules of glycine to one Fe2+ atom.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy.
2. Gestational age 14-18 weeks.
3. Mild to moderate anemia
4. No associated medical or obstetric complications.
5. Women not already receiving iron therapy.
6. Women accepted to participate in the study.

Exclusion Criteria:

1. Multiple pregnancy
2. Severe anemia
3. Iron hypersensitivity.
4. Liver diseases.
5. Women refuse to participate in the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
the rate of increase of Hemoglobin level | 8 weeks
  difference in hemoglobin concentrations before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt